CLINICAL TRIAL: NCT03022214
Title: ADAPT: Efficacy of a Dietary Supplement to Increase Resilience and Inhibit the Oxidative Stress Response During and After Exercise
Brief Title: ADAPT: Efficacy of a Dietary Supplement During and After Exercise
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Bdr2017-1
Record Dates: First submitted 2017-01-10; First posted 2017-01-16 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Dietary Supplementation During Exercise
Keywords: Dietary supplementation; Exercise; Increase Resilience; Oxidative Stress; Efficacy
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental): 5 capsules of placebo (microcrystalline cellulose) taken once in the morning with breakfast and once in the evening with dinner for two days prior to the study supervised exercise period and then one dose taken on the morning of the exercise test with the first meal
  Interventions: Dietary Supplement: Placebo
- Intervention (Experimental): For presentation to volunteers, the daily capsules will be divided into two servings, one serving to be taken in the morning with breakfast, and one serving to be taken in the evening with dinner. Each serving containing 5 capsules, as follows:
  * EnduraCell broccoli sprout powder: 3 capsules
  * Bulk Powders Green tea extract: 1 capsule
  * Bulk Powders Cinnamon Bark Extract: 1 capsule to be taken for two days prior to the study supervised exercise period and then one dose taken on the morning of the exercise test with the first meal
  Interventions: Dietary Supplement: Intervention

INTERVENTIONS:
Dietary Supplement: Placebo — Microcrystalline cellulose capsules x 5 morning and night with meals for two days prior to exercise test and 5 capsules taken on the morning of the test with the first meal
  Arms: Placebo
Dietary Supplement: Intervention — Daily capsules will be divided into two servings, one serving to be taken in the morning with breakfast, and one serving to be taken in the evening with dinner. Each serving containing 5 capsules, as follows:
  * EnduraCell broccoli sprout powder: 3 capsules
  * Bulk Powders Green tea extract: 1 capsule
  * Bulk Powders Cinnamon Bark Extract: 1 capsule taken for two days prior to exercise test and 5 capsules taken on the morning of the test with the first meal
  Arms: Intervention

SUMMARY:
Since 1948, health has been defined as "a state of complete physical, mental and social well-being, and not merely the absence of disease and infirmity" . However, a growing school of thought suggests that health represents an ability to be adaptable and flexible in response to daily stressors. It has been proposed that instead, the view of health should be "towards the ability to adapt and self-manage in the face of social, physical and emotional challenges", which has been termed "resilience".

The theory of "resilience" relates health to the body's capacity to manage daily stressors (such as physical activity or oxidative fluctuations) that challenge homeostasis, with the return to homeostasis resulting from several physiological stress responses. Although this is an all-encompassing model, and the effects of pathogens and other stress factors are also relevant, this study will centre on the physiological aspects on this theory, focussing on the disruption through exercise.

DETAILED DESCRIPTION:
The Nrf-2 pathway is the major cellular defence against oxidative and electrophilic stresses. Briefly, following dissociation from Keap1 (a scaffolding protein which binds Nrf2 and Cul3 ubiquitin ligase for proteasome degradation), Nrf-2 accumulates in the nucleus where it activates the antioxidant response element (ARE) in the promoter region of many antioxidant genes, including catalase, glutathione peroxidases (GPX), and superoxide dismutase (SOD). As such, it is an attractive target for both dietary and pharmacological interventions aiming to increase resilience to oxidative stress. Most diet-derived bioactive Nrf-2 inducers contain Michael acceptor groups (an α, β-unsaturated carbonyl moiety). Curcumin, for example, contains two Michael acceptor groups and is a known activator of Nrf-2. An additional bioactive with a Michael accepter group is trans-cinnamaldehyde (CA) (a component found in the stem bark of Cinnamomum cassia), which, like curcumin, is an Nrf-2 activator in a dose-dependent manner.

Therefore, the purpose of this study will be to assess the effect of bioactive Nrf-2 inducers, based on the presence of an α, β-unsaturated carbonyl moiety, on resilience markers such as antioxidant enzyme activities and markers of oxidative stress, such as TBARS, to an exercise challenge. The hypothesis is that specific plant bioactive increase the production of antioxidant enzyme activities at baseline, and thereby decrease levels of TBARS upon an exercise challenge. Ultimately, the use of novel resilience markers and signatures could significantly improve the ability to prove the efficacy by which pro-oxidant dietary bioactive improve lifelong health, as well as targeting those with lowest resilience as a way to make best use of limited healthcare resources.

The intervention supplement will consist of a mix of dietary bioactive with an α, β-unsaturated carbonyl moiety (provided in individual capsules), of which the efficacy to beneficially affect platelet activity, with and without a H2O2 (Hydrogen Peroxide) challenge, was recently established: sulforaphane (SUL), green tea extract (epigallocatechin gallate) (EGCG) and cinnamaldehyde (Cin).

It is intended to use a mix of dietary bioactive for the proposed human intervention study, as different compounds could affect multiple pathways and therefore, have a broader efficacy. In addition, bioavailability of compounds may be influenced by presence of other compounds, as has been suggested in the literature (effect of piperine on EGCG bioavailability).

Bioavailability data for each of these compounds were extracted from the literature and these have been used, alongside practical considerations, to decide on the dosing strategy. The desired composition of the supplement mix has been set as follows:

* SUL: ~ 14mg
* EGCG: ~ 400mg
* CIN: ~ 15mg These daily intakes should be sufficient to achieve micromolar quantities in blood plasma for between 1 and 6 hours after ingestion, and perhaps longer. .

Suitable food ingredients which can be used in the study to achieve these intakes have been sourced from reputable suppliers. These ingredients will be used to give desired intakes as follows:

* EnduraCell broccoli sprout powder (with added myrosinase): 1.5g (sufficient to provide ~ 45mg glucoraphanin, the precursor to SUL, which should release approximately ~14mg SUL).
* Bulk Powders Green tea extract: ~ 900mg (containing approximately 400mg EGCG).
* Bulk Powders Cinnamon Bark Extract: 0.75g (containing ~15 - 20mg Cin).

Due to envisaged difficulties with palatability, the ingredient mix will be encapsulated. While one of the ingredients (green tea extract) is available pre-encapsulated from the supplier, it is preferred to obtain all ingredients as free powder, and encapsulate them into size 00 capsules at Science in Sport. This will avoid difficulties with placebo blinding, as the capsules can all be given a similar appearance. Tests indicate that daily doses of cinnamon bark extract and of green tea extract will be represented by 2 capsules, each containing 375mg (cinnamon bark extract) and 450mg (green tea extract), while a daily dose of broccoli sprout powder will be represented by 6 capsules containing 250mg each. Placebo capsules will be prepared using food grade microcrystalline cellulose. Microbial testing will be carried out on all supplements.

For presentation to volunteers, the daily capsules will be divided into two servings, one serving to be taken in the morning with breakfast, and one serving to be taken in the evening with dinner. Each serving containing 5 capsules, as follows:

* EnduraCell broccoli sprout powder: 3 capsules
* Bulk Powders Green tea extract: 1 capsule
* Bulk Powders Cinnamon Bark Extract: 1 capsule

One serving of the placebo intervention contains:

• Placebo (microcrystalline cellulose): 5 capsules

Volunteers will take 5 servings just prior to the exercise challenge tests as follows:

Day -2: two servings (one in the morning and one in the evening) Day -1: two servings (one in the morning and one in the evening) Day 0: one serving (one in the morning with the first meal)

Each serving of capsules will be individually bagged and labelled with a unique identifier. Volunteers will be instructed to take a serving of capsules twice per day, with a small volume of water. They will be asked to record the unique identifier of each capsule serving after consumption, along with the time at which it was consumed. Compliance will be monitored via this daily supplement log, as well as by measuring plasma SUL metabolites.

Volunteers will be encouraged to minimise, as far as is possible, a high intake of products rich in sulforaphane (cruciferous vegetables such as Brussels sprouts, broccoli, cabbage, cauliflower, bok choy, kale, collards, broccoli sprouts, chinese broccoli, broccoli raab, kohlrabi, mustard, turnip, radish, rocket), epigallocatechin gallate (green tea) and cinnamaldehyde (cinnamon), during the 2.5 days prior to the challenge test days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, recreationally active men and women aged 18-25 BMI 18.5-30
* Healthy, recreationally active men and women aged 50-75 BMI 18.5-30

Exclusion Criteria:

* Physician diagnosed diabetes or chronic disease including asthma
* Pregnancy
* Uncontrolled Hypertension
* Musculo-skeletal problems
* Use of some dietary supplements (e.g. antioxidants, fish oils, vitamins_
* Taking of prescription medicines
* In the 18-25 group, Physical Activity levels below moderate (Moderate = greater than 2.5 and less than 5.0 hrs /week including 0.5-1.5 hr/week moderate to intense exercise)
* In the 50-75 group, activity levels below the minimal recommendations for daily physical activity (less than 30 min/day, 5 days/week)
* Participation in another research study
* Not being able to speak or understand English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Markers of Oxidative Stress | 18months
  Plasma TBARS:Plasma TBARS will be measured by HPLC (High Performance Liquid Chromatography).

SECONDARY OUTCOMES:
Antioxidant enzyme activity | 18months
  Glutathione peroxidase, superoxide dismutase, and acetaldehyde dehydrogenase will be measured in plasma by spectrophotometer.
Marker of Oxidative Stress | 18months
  Plasma F2-Isoprostanes: will be measured by ELISA.
Markers of Inflammation | 18months
  Plasma high sensitivity C-Reactive Protein (hs-CRP): Plasma hsCRP will be assessed by automated analysis using KONE.
Plasma Interleukin-6 (IL-6) | 18months
  Plasma IL-6 will be assessed by ELISA.
Plasma Tumour-Necrosis Factor - alpha (TNF-α) | 18months
  Will be assessed by ELISA.
Metabolic risk markers | 18months
  Plasma insulin: Plasma insulin will be assessed by ELISA.
Plasma glucose | 18months
  Plasma glucose will be assessed by automated analysis using KONE.
Plasma non-esterified fatty acids (NEFA) | 18months
  Will be measured by automated analysis using KONE.
Markers of muscle damage | 18 months
  Plasma Creatine Kinase activity will assessed by spectrophotometer Plasma Lactate dehydrogenase activity will assessed by spectrophotometer
Markers of platelet function | 18 months
  Thrombin generation
Counter Movement Jump | 18months
  This is a test of lower body strength and will be assessed throughout the study visits using a vertical jump meter.
Subjective Ratings | 18months
  Questionnaires to be applied during exercise challenge test days
Wellness Questionnaire | 18months
  To assess lifestyle factors such as fatigue, sleep, and mood.
Perceived Soreness of quadriceps | 18months
  Rating of perceived soreness (pre, post, 48hr post) - Volunteers will rate their perceived soreness in their quadriceps on a ten point scale.
Perceived Exhaustion | 18months
  Ratings of perceived exhaustion (during exercise challenge) - Volunteers will rate their perceived exhaustion using Borg's modified R.P.E scale (10 point).

CONTACTS AND LOCATIONS:
Overall Officials: Baukje De Roos, Msc, PhD, Principal Investigator — The Rowett Institute, University of Aberdeen, Foresterhill, Aberdeen, AB25 2ZD
Locations (1):
- University of Aberdeen, The Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No